CLINICAL TRIAL: NCT05149456
Title: Study of the Prevalence of Peripheral Artery Occlusive Disease (PAOD) in Women Hospitalized for Type 1 Myocardial Infarction in Intensive Cardiology Care
Brief Title: Peripheral Artery Occlusive Disease (PAOD) in Women Hospitalized for Type 1 Myocardial Infarction in Intensive Cardiology Care
Acronym: AOMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8373
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: PAOD - Peripheral Arterial Occlusive Disease
Keywords: Peripheral Arterial Occlusive Disease; PAOD; Cardiovascular risk factors; Myocardial infarction
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The cardiovascular risk of women has been the subject of particular interest in recent years, in the world, in particular under the impetus of Cardiology companies, with more and more work focusing on the specificities of these diseases in women as well as differences in terms of management and prognosis with a literature mainly based on American data and which focuses particularly on ischemic heart disease.

The expected results are to have a prevalence of PAOD in an Alsatian cohort, most of the data we currently have from American data, with analysis of the impact of specific and non-specific risk factors in this cohort and their weight in PAOD.

ELIGIBILITY:
Inclusion criteria:

* Adult woman (≥18 years old)
* Patient hospitalized in an Intensive Cardiology Unit (ICU) at the HUS for a type 1 myocardial infarction confirmed according to the criteria of the fourth universal definition of the ESC between 01/01/2021 to 30/06/2021 inclusive
* Patient who did not express her opposition to the reuse of her data for scientific research purposes.

Exclusion criteria:

* Patient who expressed her opposition to participating in the study
* Impossibility of providing the subject with enlightened information (difficulties in understanding the subject, MMS <20/30…)
* Non-type 1 or unconfirmed myocardial infarction
* Unstable or refractory shock state at the time of the echodoppler examination
* Complication of the coronary angiography approach, in the case of femoral approach only, requiring surgical management.
* Patient under curatorship, guardianship or judicial safeguard.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult woman hospitalized in an Intensive Cardiology Unit (ICU) at the HUS for a type 1 myocardial infarction confirmed according to the criteria of the fourth universal definition of the ESC between 01/01/2021 to 30/06/2021 inclusive
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Study of the prevalence of peripheral artery occlusive disease (PAOD) | Files analysed retrospectively from January 01, 2021 to Jun 30, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Dominique STEPHAN, MD, PhD, Principal Investigator — Service des Maladies VASC-HTA-Pharmacologie Clinique - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service des Maladies VASC-HTA-Pharmacologie Clinique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France